CLINICAL TRIAL: NCT01181648
Title: Surviving Oropharynx Cancer: Long-Term Impact of Human Papillomavirus (HPV) on Quality of Life
Brief Title: Long-Term Impact of Human Papillomavirus (HPV) on Quality of Life
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 10-111
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Squamous Cell Carcinoma of the Oropharynx
Keywords: Survivor; Human Papillomavirus (HPV); Quality of Life; Surviving Oropharynx Cancer; 10-111
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- oropharynx cancer survivors: This study has two components. First, we will conduct a cross-sectional survey of 200 oropharynx cancer survivors, diagnosed with HPV+ tumors, who are at least 12 months from their last treatment. Second, in a subset of 20 survivors of HPV+ oropharynx cancer, we will conduct in-depth, semi-structured, face-to-face interviews addressing the psychosocial impact of the HPV diagnosis.
  Interventions: Behavioral: questionnaire and semi-structured interviews

INTERVENTIONS:
Behavioral: questionnaire and semi-structured interviews — Survivors will be asked to complete a brief, self-administered, paper-based survey to assess quality of life, mental health and employment status following completion of therapy. Second, in a subset of 20 survivors of HPV+ oropharynx cancer, we will conduct in-depth, semi-structured, face-to-face interviews addressing the psychosocial impact of the HPV diagnosis. A follow up letter will be sent to participants who do not return their completed study questionnaires.

SUMMARY:
The investigators are doing this study to learn about the quality of life patients have at the end of treatment. Some patients' cancers are related to human papilloma virus or HPV; others are not. HPV is a virus that can be sexually transmitted and is known to cause some types of cancers. If your throat cancer was related to HPV, your doctor can discuss this with you in detail. The investigators want to see if there are differences in quality of life between patients whose cancers are caused by HPV and those who cancers are not caused by HPV. Throat cancers caused by HPV behave differently than throat cancers not caused by HPV. The investigators believe that patients with these two different types of throat cancer will also have different experiences after completing therapy. The investigators would like to understand what those differences are. The long-term goal of this study is to see what symptoms most patients have. The investigators can then try to treat them earlier, and hopefully, improve the symptoms. The investigators will also be able to plan more research to improve treatment for symptoms following treatment for cancer of the mouth and throat.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of squamous cell carcinoma of the oropharynx confirmed by the pathology department at MSKCC
* Completed last treatment for oropharynx cancer (surgery, chemotherapy, or radiation) at least 12 months and no more than 5 years before the date of study enrollment
* Known tumor status or tumor available for HPV testing [based on chromogenic in situ hybridization with wide spectrum HPV probe (HPV III family 16 probe (Ventana) with affinity to HPV genotypes 16, 18, 31, 33, 35, 45, 51, 52, 56, 58, and 66) or p16 immunohistochemistry done in a Clinical Laboratory Improvement Amendment (CLIA)-approved laboratory; if either of these 2 tests are positive, the patient is classified as positive].
* Able to speak and read English (study questionnaire-Aim 1 and interview guide-Aim 2 are currently only available in English).
* Received at least one component of treatment for oropharynx cancer at MSKCC or the regional network sites
* If radiation therapy was part of treatment, it must have been delivered at MSKCC or the regional network sites
* For Aim 2 only, diagnosed with an HPV+ oropharynx cancer and have knowledge of this diagnosis prior to study enrollment

Exclusion Criteria:

* Diagnosed with recurrent disease following completion of primary curative treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified through a Dataline query. While Dataline should capture most eligible patients, potential subjects can also be identified by a member of the Head and Neck DMT.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2010-08; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
To assess quality of life in survivors | 2 years
  of oropharynx cancer at least one year after completion of curative treatment in patients with HPV+ disease versus HPV- disease.

SECONDARY OUTCOMES:
Explore the psychosocial impact of a HPV diagnosis | 2 years
  on survivors of HPV+ oropharynx cancer

CONTACTS AND LOCATIONS:
Overall Officials: Shrujal Baxi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center at Phelps, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm